CLINICAL TRIAL: NCT03868514
Title: "PRO-Pocket" - International Prospective Multicenter Post Market Clinical Follow Up to "Patient Reported Outcome" in Primary or Secondary Breast Reconstruction After Mastectomy Using a Titanised Polypropylene Mesh (TiLOOP® Bra Pocket)
Brief Title: Post Market Clinical Follow Up to "Patient Reported Outcome" Using a Titanised Polypropylene Mesh (TiLOOP® Bra Pocket)
Acronym: PRO-Pocket
Status: Completed | Type: Observational
Sponsor: pfm medical gmbh (Industry)
Responsible Party: Sponsor
Other Study IDs: P050001 TiLOOP® Bra Pocket
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Breast Reconstruction After Mastectomy; Breast Neoplasm; Breast Cancer; Breast Diseases
Keywords: breast reconstruction; surgical mesh; synthetic mesh; patient reported outcome; breast cancer; mesh
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TiLOOP Bra Pocket: Medical Device
  Interventions: Device: TiLOOP® Bra Pocket

INTERVENTIONS:
Device: TiLOOP® Bra Pocket — Primary or secondary breast reconstruction following mastectomy with titanised polypropylene mesh TiLOOP® Bra Pocket

SUMMARY:
"PRO-Pocket" - International prospective multicentre Post Market Clinical Follow Up to "Patient reported outcome" in primary or secondary breast reconstruction after mastectomy using a titanised polypropylene mesh (TiLOOP® Bra Pocket)

DETAILED DESCRIPTION:
This international, multicentre, non-randomised, observational clinical device investigation will be performed to obtain post market information on TiLOOP® Bra Pocket surgical meshes for a period of up to two years. In particular, on patient reported satisfaction (BreastQTM), cosmetic outcome and the rate of complications.

The objective of the clinical Investigation is to establish the efficacy and safety of the TiLOOP® Bra Pocket.

The Investigation will be performed in ten clinical centres in Germany and Austria.

ELIGIBILITY:
Inclusion Criteria:

Age [≥ 18]

Indications of breast reconstruction: histologically confirmed breast cancer, precancerous lesions (DCIS, LCIS), mutation carrier with increased breast cancer risk, strong family history (lifetime risk > 15%)

The patient is capable to realise the nature, aims and possible consequences of the clinical trial (MPG §20.2.1)

Patient information has been provided and all written consents of the patient are available

Exclusion Criteria:

Metastatic breast cancer

Patient with known contraindications against mesh-assisted or plastic-reconstructive breast surgery according to the instruction for use

Patient is kept in an institution under judicial or official orders (MPG §20.3)

Participate in another operative clinical trial, if it relates to the area of reconstructive breast surgery and/or influences the primary endpoint of the clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with indicated implant based breast reconstruction after mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Quality of Life - Patient reported outcome | 12 months after study treatment
  The primary endpoint is defined as the change of the four BreastQ domain scores before study treatment compared to twelve months after study treatment. The BreastQ questionnaire yields a domain score in the range from zero to 100. Wheras a score of 100 is the best score. The study hypothesis is that the patient's QoL after the study intervention treatment is not worse than the QoL prior to the intervention study treatment . The following four domains are relavant: Satisfaction with breasts, Psychosocial well-being, Physical well-being:chest and Sexual well-being.

SECONDARY OUTCOMES:
Quality of Life - Patient reported outcome | 6 and 24 months after study treatment
  The change of the four BreastQ domain scores before study treatment compared to six months and 24 months after study treamtment.
Complication rate | 6, 12 and 24 months after study treatment
  The number and rate of occurrence of adverse events is reported as a secondary endpoint along with a tabulation of the types of adverse events (6, 12 and 24 months after study treatment).
Cosmetic outcome | 6, 12 and 24 months after study treatment
  The cosmetic outcome is assessed based on photographs 6, 12 and 24 months after study treatment by descriptive statistics (an independent expert, the physician in charge and the patient assess the cosmetic outcome).

CONTACTS AND LOCATIONS:
Locations (12):
- Universitätsklinik für Frauenheilkunde, Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Germany (11):
  - Vivantes Klinikum Am Urban, Berlin
  - DRK Kliniken Westend, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Kliniken Essen Mitte; Evang. Huyssens-Stiftung, Essen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Heidelberg, Heidelberg
  - Rotkreuzklinikum München, Munich
  - Klinikum rechts der Isar der Technischen Universität München, Munich
  - Universitätsklinikum Ulm, Ulm
  - GRN Klinik Weinheim, Weinheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: pfm medical study information — https://www.pfmmedical.com/knowledge/studies/study_on_tiloop_bra_pocket/index.html